CLINICAL TRIAL: NCT06590974
Title: Special Drug Use Surveillance Study of Ceprotin for Intravenous Injection 1000IU (All-Case Surveillance)
Brief Title: A Study of Freeze-dried Human Protein C Concentrate (TAK-662) in Participants With Congenital Protein C Deficiency
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-662-4002; jRCT2031240322 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Protein C Deficiency
Keywords: Ceprotin/Protein C Deficiency
MeSH Terms: conditions — Protein C Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Freeze-dried Human Protein C Concentrate (TAK-662): Participants will be administered Freeze-dried Human Protein C Concentrate (TAK-662) intravenous injection.
  Interventions: Drug: Freeze-dried Human Protein C Concentrate

INTERVENTIONS:
Drug: Freeze-dried Human Protein C Concentrate — Freeze-dried Human Protein C Concentrate (TAK-662) intravenous injection

SUMMARY:
This study is conducted in Japan of Freeze-dried Human Protein C Concentrate (TAK-662) used to treat participants with congenital protein C deficiency.

The main aim of the study is to evaluate for adverse events and effectiveness of congenital protein C deficiency (TAK-662).

During the study, participants with congenital protein C deficiency will be administered with TAK-662 intravenous injection in under routine normal practice. The investigators will evaluate adverse events due to TAK-662 for 12 months. For participants who will be administered in long-term supplementation of TAK-662 after acute treatment or short-term supplementation, the investigator will evaluate for 24 months as a maximum. The study sponsor will not be involved in how the participants are administered but will be recorded what happens during the study.

ELIGIBILITY:
Inclusion Criteria:

- All participants with congenital protein C deficiency who are administered with Freeze-dried Human Protein C Concentrate (TAK-662).

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this study are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience at Least One Treatment-Emergent Adverse Events (TEAE) | Up to 12 months (For participants who will be administered in long-term supplementation of TAK-662 after acute treatment or short-term supplementation, up to 24 months as a maximum)

SECONDARY OUTCOMES:
Number of Participants who Experience at Least One TEAE of Venous Thromboembolism | Up to 12 months (For participants who will be administered in long-term supplementation of TAK-662 after acute treatment or short-term supplementation, up to 24 months as a maximum)
Number of Participants who Experience at Least One TEAE of Purpura Fulminans | Up to 12 months (For participants who will be administered in long-term supplementation of TAK-662 after acute treatment or short-term supplementation, up to 24 months as a maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).